CLINICAL TRIAL: NCT04678817
Title: A Prospective Observational Study of Preference for and Efficacy of Oral Levonorgestrel Emergency Contraception With Same Day Etonogestrel Contraceptive Implant Compared to Established Pregnancy Rates With Oral Levonorgestrel Emergency Contraception Alone
Brief Title: Same Day Oral EC and Implant Initiation
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 137011
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Contraception
Keywords: emergency contraception; contraceptive implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Etonogestrel contraceptive implant with oral levonorgestrel: Participants who select the Etonogestrel implant with oral levonorgestrel for emergency contraception
  Interventions: Device: Etonogestrel contraceptive implant with oral levonorgestrel
- Levonorgestrel intrauterine device: Participants who select the levonorgestrel intrauterine device for emergency contraception
  Interventions: Device: Levonorgestrel intrauterine device
- Copper T380A intrauterine device: Participants who select the Copper T380A intrauterine device for emergency contraception
  Interventions: Device: Copper T380A intrauterine device

INTERVENTIONS:
Device: Etonogestrel contraceptive implant with oral levonorgestrel — Participants who present for emergency contraception and select the Etonogestrel contraceptive implant with oral levonorgestrel
  Groups: Etonogestrel contraceptive implant with oral levonorgestrel
Device: Levonorgestrel intrauterine device — Participants who present for emergency contraception and select the Levonorgestrel intrauterine device
  Groups: Levonorgestrel intrauterine device
Device: Copper T380A intrauterine device — Participants who present for emergency contraception and select the Copper T380A intrauterine device
  Groups: Copper T380A intrauterine device

SUMMARY:
This is a study for clients presenting for emergency contraception (EC). EC is used to prevent pregnancy after unprotected intercourse. Clients presenting for EC may be offered either the copper or hormonal IUD or oral EC. Current guidelines allow for same-day implant initiation at the time of an EC encounter, as long as oral LNG EC is co-administered. This study will look at pregnancy rates and clients willingness to receive same-day implant + oral EC and same-day IUDs.

DETAILED DESCRIPTION:
Recommended options for EC include oral EC (levonorgestrel (LNG), ulipristal acetate (UPA), or combination oral contraceptive pills), or the copper intrauterine device (IUD). Recent data will also allow women presenting for EC to be offered the LNG IUD. These recommendations leave out the only other long-acting reversible contraceptive (LARC), the ENG implant. Current guidelines allow for same-day ENG implant initiation at the time of an EC encounter, as long as oral LNG EC is co-administered. We lack data on pregnancy risk for the EC-eligible population desiring same-day ENG implant placement and oral EC.

Women presenting for EC often need ongoing contraception, but clinical practice is not standardized in same-day counseling and initiation due to system, provider, and client-level barriers. Interest in LARC use continues to increase as well as same-day contraception initiation at the time of an EC encounter. Women presenting for EC may not have considered LARC options before. Generating estimates and continuation rates for same-day initiation with an EC encounter will improve contraceptive options for women seeking EC.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Age 18-35 years
* Fluent in English and/or Spanish
* BMI < 30 kg/m2
* No known contraindication to either the ENG contraceptive implant or oral LNG EC using the CDC Medical Eligibility Criteria for Contraceptive Use 2016
* Negative urine pregnancy test
* Willing to abstain from further UPI in the 7 days following insertion
* Know the date of their last menstrual period
* Regular menstrual cycle (24-35 days)
* Be willing to comply with the study requirements
* Desiring to avoid pregnancy for at least 12 months

Exclusion Criteria:

* Current pregnancy or breastfeeding
* Previous use of oral EC in the current cycle
* Report of UPI beyond 5 days in current cycle
* Vaginal bleeding of unknown etiology
* Allergy to LNG or ENG, IUD or implant in-place
* History of permanent contraception through sterilization or hysterectomy
* Monogamous partner with a vasectomy
* Depo-provera injection within past 15 weeks

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study population will be recruited from participating Planned Parenthood of Utah clinics.
Sampling Method: Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Gawron, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Planned Parenthood Association of Utah, Salt Lake City, Utah
  - Planned Parenthood Association of Utah, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to share with other researchers.

REFERENCES:
- [Derived] Carter G, Pangasa M, Sexsmith CD, Elliott S, Turok DK, Gawron LM. Selection of long acting reversible contraception methods by emergency contraception clients: A prospective observational study. Contraception. 2025 Jan;141:110701. doi: 10.1016/j.contraception.2024.110701. Epub 2024 Sep 4. PMID 39241904
- [Derived] Gawron LM, Sexsmith CD, Carter G, Kaiser JE, Pangasa M, Turok DK. Efficacy of oral levonorgestrel emergency contraception with same day etonogestrel contraceptive implant: A prospective observational study. Contraception. 2024 Mar;131:110344. doi: 10.1016/j.contraception.2023.110344. Epub 2023 Nov 25. PMID 38008305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Emergency contraception clients age 18-35y at four Utah family planning clinics between February 2021 and April 2023 received information about oral emergency contraception and three long acting reversible contraception options: the etonogestrel implant with same-day oral levonogestrel, the 52mf levonogestrel intrauterine device, and the copper T380A intrauterine device.
Pre-assignment Details: We excluded nine potential participants for long acting reversible contraception contraindications and another four due to failed intrauterine device insertions
Period: Overall Study
Arm/Group | Etonogestrel Contraceptive Implant With Oral Levonorgestrel | Levonorgestrel Intrauterine Device | Copper T380A Intrauterine Device
Started | 160 | 61 | 72
Completed | 132 | 61 | 72
Not Completed | 28 | 0 | 0
Not completed — Lost to Follow-up | 28 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etonogestrel Contraceptive Implant With Oral Levonorgestrel | Levonorgestrel Intrauterine Device | Copper T380A Intrauterine Device | Total
Number analyzed (Participants) | 160 | 61 | 72 | 293
Age, Customized [Count of Participants; unit: Participants]
  <20 years | 41 | 8 | 10 | 59
  20-24 years | 72 | 30 | 28 | 130
  25-29 years | 24 | 9 | 15 | 48
  30+ years | 23 | 14 | 19 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 61 | 72 | 293
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black/ African American | 9 | 2 | 2 | 13
  Hispanic/ Latina | 80 | 15 | 16 | 111
  Race not listed | 14 | 5 | 2 | 21
  White | 57 | 39 | 52 | 148
Region of Enrollment [Number; unit: participants]
  United States | 160 | 61 | 72 | 293
Body mass index [Count of Participants; unit: Participants]
  < 25 kg/m2 | 71 | 30 | 47 | 148
  25 - 29.9 kg/m2 | 36 | 18 | 15 | 69
  30+ kg/m2 | 53 | 12 | 9 | 74
  missing | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rate at One-month
Description: To determine a point estimate for the one-month pregnancy rate following guideline supported same-day initiation of an etonogestrel (ENG) implant plus oral levonorgestrel (LNG) emergency contraception (EC).
Time Frame: one month
Population: Participants who selected the Etonogestrel contraceptive implant with oral levonorgestrel for emergency contraception reported pregnancy test results at 1 month post enrollment. Participants who selected a Levonorgestrel Intrauterine Device or a Copper T380A Intrauterine Device only completed an enrollment survey and were not followed for longitudinal outcomes.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Etonogestrel Contraceptive Implant With Oral Levonorgestrel: Participants who selected the Etonogestrel contraceptive implant with oral levonorgestrel for emergency contraception
Arm/Group | Etonogestrel Contraceptive Implant With Oral Levonorgestrel
Number analyzed (Participants) | 153
percentage of participants | 1.96 [0.51 to 6.07]

2. Primary Outcome: Comparing Proportions of EC Clients Desiring ENG Implant With Oral EC vs IUD
Description: To determine the proportion of EC clients willing to initiate a same-day ENG implant with oral LNG EC compared to same-day initiation of intrauterine devices for EC.
Time Frame: 2 years
Population: Number of participants choosing each method out of total 293 enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Etonogestrel Contraceptive Implant With Oral Levonorgestrel | Levonorgestrel Intrauterine Device | Copper T380A Intrauterine Device
Number analyzed (Participants) | 160 | 61 | 72
percentage of participants | 54.6 | 20.8 | 24.6

3. Secondary Outcome: Continuation Rate
Description: 12-month continuation rate of the ENG implant with same-day initiation at an EC encounter.
Time Frame: 12 months
Population: Number of participants from Arm 1 who selected an etonogestrel implant and completed a 12 month follow up survey. The outcome measure below is the percentage who reported implant continuation at 12 months. Participants who selected a Levonorgestrel Intrauterine Device or a Copper T380A Intrauterine Device only completed an enrollment survey and were not followed for longitudinal outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Etonogestrel Contraceptive Implant With Oral Levonorgestrel
Number analyzed (Participants) | 132
Participants | 79

4. Secondary Outcome: Discontinuation Rate and Reasons
Description: Rate and reasons for ENG implant discontinuation in the 12 months following same-day initiation at an EC encounter.
Time Frame: 12 months
Population: Number of participants from Arm 1 who selected an etonogestrel implant and reported discontinuation of the implant in the 12 months of follow up survey.s The outcome measures below are the percentage who reported reasons for method implant discontinuation. More than 1 reason could be selected by participants. Participants who selected a Levonorgestrel Intrauterine Device or a Copper T380A Intrauterine Device only completed an enrollment survey and were not followed for longitudinal outcomes.
Measure: Number; unit: percentage of participants
Arm/Group | Etonogestrel Contraceptive Implant With Oral Levonorgestrel
Number analyzed (Participants) | 53
percentage of participants
  Discontinued for bleeding | 51
  Discontinued for mood changes | 41
  Discontinued for weight gain | 37
  Discontinued for bloating | 24
  Discontinued for cramping | 20

ADVERSE EVENTS:
Time Frame: 30 days post enrollment
Arm/Group | Etonogestrel Contraceptive Implant With Oral Levonorgestrel | Levonorgestrel Intrauterine Device | Copper T380A Intrauterine Device
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/61 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/160 | 0/61 | 0/72
Other Adverse Events (participants affected / at risk) | 0/160 | 0/61 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT04678817/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT04678817/ICF_000.pdf